CLINICAL TRIAL: NCT03432624
Title: A Clinical Validation Study on the Efficacy of MicroRNA-25 Level Detection in Assisting the Diagnosis of Pancreatic Cancer
Brief Title: Detection of MicroRNA-25 in the Diagnosis of Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Director, Head of Otolaryngology, Principal Investigator, Clinical Professor, Fudan University
Other Study IDs: CSPAC-030
Record Dates: First submitted 2018-01-24; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Carcinoma, Pancreatic Ductal
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Experiment Subgroup, Group One: Experiment Subgroup, Group One consists of pancreatic cancer patients, in which 120 are operable, and 120 are not operable.
  Interventions: Diagnostic Test: Serum MicroRNA-25 detection
- Control Subgroup, Group One: Control Subgroup, Group One consists of 150 patients, in which 30 are of gallbladder carcinoma, 60 are of biliary tract lower segment carcinoma, 60 are of gastrointestinal carcinoma.
  Interventions: Diagnostic Test: Serum MicroRNA-25 detection
- Interference Subgroup, Group One: Interference Subgroup, Group One consists of 150 patients, in which 60 are of chronic pancreatitis, 90 are of other types of pancreatic tumor, in which 30 are of IPMN (intraductal papillary mucinous neoplasm), 30 are of SPT (solid pseudopapillary tumor of pancreas), and 30 pancreatic cystic adenoma.
  Interventions: Diagnostic Test: Serum MicroRNA-25 detection
- Experiment Subgroup, Group Two: Group Two consists of 210 patients selected from Group One, of which the Experiment Subgroup, Group Two consists of the 120 operable pancreatic cancer patients who have had successful surgery.
  Interventions: Diagnostic Test: Serum MicroRNA-25 detection
- Control Subgroup, Group Two: Control Subgroup, Group Two consists of 90 patients of other cancers who have had successful surgery, in which 30 are of gallbladder carcinoma, and 60 are of biliary tract lower segment carcinoma.
  Interventions: Diagnostic Test: Serum MicroRNA-25 detection

INTERVENTIONS:
Diagnostic Test: Serum MicroRNA-25 detection — The level of microRNA-25 in serum of patients will be detected using the MicroRNA (microRNA-25) Qualitative Detection Kit (Fluorescent PCR Method) and following the manufacture's instruction.*all arms are given the same intervention.

SUMMARY:
Pancreatic cancer represents the most lethal of the common malignancies, with a 5-year survival rate of less than 5%. For patients who, when are diagnosed of pancreatic cancer, are eligible for potentially curative resection, the mortality and morbidity rates after surgery can improve significantly, but who accounts for no more than 20% of all pancreatic patients. It is therefore an effective way to improve the treatment efficacy for pancreatic cancer by discovering novel detection methods for pancreatic cancer, especially at early stages. MicroRNAs have been proved in recent years as functional disease markers, and circulating microRNA-25 is reported of high pancreatic cancer specificity and can be used as a novel marker for pancreatic cancer. A detection kit "MicroRNA (microRNA-25) Qualitative Detection Kit (Fluorescent PCR Method)" is produced and proven to be effective in assisting the diagnosis of pancreatic cancer through clinical trials held independently in three state-level hospitals in China. To further validate the efficacy of the kit, the researchers in this study intend to compare the sensibility and specificity of microRNA-25 level detection and other diagnosis methods, including detection of conventional tumor markers (CA19-9, CA125, CA50, CEA) and imaging (CT, MRI, PET/CT), both in separation and combined, in the diagnosis of pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer (mainly pancreatic ductal adenocarcinoma, PDAC) is a disease with extremely poor prognosis, and is often fatal. Surgical resection is the only potentially curative technique for management of PDAC, but only approximately 15% to 20% of patients are candidates for pancreatectomy at the time of diagnosis. For these patients, however, the mortality and morbidity rates after surgery can improve significantly. It is therefore an effective way to improve the treatment efficacy for pancreatic cancer by discovering novel detection methods for pancreatic cancer, especially at early stages.

MicroRNAs are a type of non-encoding single-stranded small RNAs with a length of ~22nt. They can regulate the expression of their target mRNAs by inhibiting their translation into proteins. MicroRNAs participate in all physiological and pathological activities, and their abnormal expression profiles are proven to be closely related to the occurrence and development of diseases, including cancer. Recent studies have further proved that not only tissue/cell-line based microRNAs, but circulating microRNAs can be stably detected, and their expression profiles can function as novel markers to be used in the diagnosis and prognosis of diseases.

Pancreatic cancer specific microRNA profiles have also been reported, amongst which microRNA-25 is found to be significantly upregulated in pancreatic cancer patients. There are also studies try to improve the efficacy of pancreatic cancer diagnosis by combining detection of microRNA and CA19-9. Further are there studies proving microRNA-25 as a highly potential marker for pancreatic cancer. A detection kit "MicroRNA (microRNA-25) Qualitative Detection Kit (Fluorescent PCR Method)" is produced and proven to be effective in assisting the diagnosis of pancreatic cancer through clinical trials held independently in three state-level hospitals in China.

To further validate the efficacy of the kit, the researchers in this study intend to compare the sensibility and specificity of microRNA-25 level detection and other diagnosis methods, including detection of conventional tumor markers (CA19-9, CA125, CA50, CEA) and imaging (CT, MRI, PET/CT), both in separation and combined, with Cohort One in the diagnosis of pancreatic cancer at early stages, to validate the efficacy of microRNA-25 detection in the differentiation of pancreatic cancer and other related diseases, to investigate the relation between microRNA-25 level and pancreatic staging. Patients in Group One will receive a microRNA-25 level detection at the time of diagnosis, along with conventional tumor marker detection and imaging tests, and then be confirmed by pathological study. And, to investigate the efficacy of microRNA-25 level detection in the curative efficacy evaluation and relapse monitoring, patients of Group Two (selected from Group One) will receive a microRNA-25 level detection within one month after surgery and before starting adjuvant therapy, followed by a microRNA-25 level detection every three months along with normal follow-up tests, until relapse is observed with imaging tests.

ELIGIBILITY:
Inclusion Criteria:

Group One:

1. Patient aged 18 years old and above at the time of signing the ICF.
2. Prior to blood sample withdraw, patient not treated with systematic anti-tumor therapy, including long-acting somatostatin analogues, interferons, PRRT (Peptide Receptor- Radionuclide Therapy), mTOR inhibitors and chemotherapy; not treated with radiotherapy or neo-adjuvant therapies.
3. Differences:

Experiment Subgroup: Patients diagnosed or highly-suspected of pancreatic cancer, among whom:

Operable: Patients confirmed with pancreatic cancer by pathological test, and evaluated by MDT as "operable" and "probably operable"; Not operable: Patients confirmed with pancreatic cancer by cytological test (exfoliative cytology or fine needle puncture biopsy), or highly suspected of pancreatic cancer by the MDT referring to disease history, clinical manifestations, lab test and imagining results.

Control Subgroup: Patients confirmed with gallbladder carcinoma, biliary tract lower segment carcinoma, and gastrointestinal carcinoma by pathological test.

Interference Subgroup: Patients diagnosed of chronic pancreatitis, IPMN (intraductal papillary mucinous neoplasm), SPT (solid pseudopapillary tumor of pancreas), pancreatic cystic adenoma.

Group Two:

1. Patient aged 18 years old and above at the time of signing the ICF, and with an expected survival time of over 12 months.
2. Prior to the first blood sample withdraw after surgery, patient not treated with radiotherapy or adjuvant therapy.
3. Differences:

Experiment Subgroup: Patients confirmed of pancreatic cancer and received successful curative operation.

Control Subgroup: Patients confirmed of gallbladder carcinoma and biliary tract lower segment carcinoma, and received successful curative operation.

Exclusion Criteria

Group One:

1. Patient in the period of acute infection.
2. Patient treated with therapies or drugs prior to blood withdraw.
3. Blood sample shows jaundice (TBIL≥17.1μmol/L) and hematolysis (to be decided by the serum sample preparer).
4. Blood sample has been stored for one year and above.

Group Two:

1. Patient treated with therapies or drugs prior to first blood withdraw after surgery.
2. Patient shows symptoms of remote metases.
3. Blood sample shows jaundice (TBIL≥17.1μmol/L) and hematolysis (to be decided by the serum sample preparer).
4. Blood sample has been stored for one year and above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed and treated at the Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Fourfold Table Analysis Indexes | throughout the trial, average one year
  Using the Fourfold Table to analyze the diagnosis value of the tested reagent in comparison with the golden standard (pathological test) from mainly four indexes: Sensitivity, Specificity, Total Coincidence Rate and Youden Index (%).
  Fourfold Table Tested reagent Golden standard Total Positive (D+) Negative (D-) Positive (T+) a b a+b Negative (T-) c d c+d Total a+c b+d N=a+b+c+d
  1. Sensitivity: Se=P(T+|D+)=a/(a+c)
  2. Specificity: Sp=P(T-|D-)=d/(b+d)
  3. Total Coincidence Rate: TC= (a+d)/N
  4. Youden Index: YI=Se+Sp-1

SECONDARY OUTCOMES:
Statistical Analysis Indexes | throughout the trial, average one year
  Statistical Analysis will evaluate the diagnosing efficacy of the tested reagent with two indexes, Kappa Value and AUC:
  Kappa Value (K Value) Analysis: to investigate the consistency of the tested reagent with golden standard.
  The definition of K is:
  K=(p_0-p_e)/(1-p_e ), Where p0 is the relative observed agreement of the tested reagent and/or the comparison reagents (identical to accuracy), and pe is the hypothetical probability of chance agreement, using the observed data to calculate the probabilities of each observer randomly seeing each category.
  AUC (%): to investigate the diagnosing efficacy of the tested reagent through calculating the AUC (Area Under the ROC Curve).
  The ROC curve is created by plotting the true positive rate (TPR) against the false positive rate (FPR) at various threshold setting. The TPR is also known as sensitivity. The FPR is also known as the fall-out or probability of false alarm and can be calculated as (1-specificity).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No